CLINICAL TRIAL: NCT06711796
Title: Measurement of Muscle Relaxation of the Hand in From Two Muscles and Two Hand Positions
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R23091L
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Relaxation
Keywords: Train of four; EMG

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: Patients undergiong surgery with no need for muscle relaxation
  Interventions: Device: emg measurement in adductor pollucis

INTERVENTIONS:
Device: emg measurement in adductor pollucis — EMG measurement from adductor pollucis and dorsal interosseus muscles in supination and pronation using increasing stimulation current

SUMMARY:
Does movement of hand from supination to pronation affect the cut threshold for electomyography (EMG) relaxation measurement Does the threshold level differ between adductor pollucis and dorsal interosseus muscle

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* American society of anesthesiology (ASA) classification 1-2
* Elective surgery under general anesteshia with no planned need for muscle relaxation
* Body mass index <35 kg/m3

Exclusion Criteria:

* Know central nervous system disease
* Know central nervous system impairment
* known medication affection peripheral nervous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery with estimated time over 45 minutes and no need for muscle relaxation
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
To differ the difference in the stimulation current between adductor pollucis and dorsal interosseus muscles | 30 minutes
  Defining the supramaximal stimulation current in the hand using EMG muscle rekaxation
To differ the stimulation threshold in hand supination and pronation postures | 30 minutes
  Measuring the EMG stimulation threshold in two hand postures

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
Physionet registry - pseudonymised measurement data
Supporting Information: Study Protocol, CSR
Time Frame: 1.1.2026-1.1.2030
Access Criteria: open registry
URL: https://physionet.org/about/database/